CLINICAL TRIAL: NCT01128920
Title: Reduction of Medical Complications Associated With Injection Drug Use
Brief Title: Reducing Health Problems Associated With Injection Drug Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Northern Colorado (Other)
Collaborators: University of Colorado, Denver (Other); Butler Hospital (Other)
Responsible Party: Principal Investigator, Kristina Phillips, Associate Professor, University of Northern Colorado
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DA026773-01
Record Dates: First submitted 2010-05-19; First posted 2010-05-24 (Estimated); Last update posted 2012-01-04 (Estimated); Status verified 2011-12

CONDITIONS: Intravenous Drug Abuse; HIV Infections
Keywords: bacterial infections; skin infections; HIV; Hepatitis C; risk reduction intervention
MeSH Terms: conditions — Substance Abuse, Intravenous; HIV Infections; Bacterial Infections; Cellulitis; Hepatitis C

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Skin and Needle Hygiene Intervention (Experimental)
  Interventions: Behavioral: Skin and Needle Hygiene Intervention
- Assessment-Only Condition (Experimental)
  Interventions: Other: No intervention - assessment-only condition

INTERVENTIONS:
Behavioral: Skin and Needle Hygiene Intervention — Intervention incorporates psychoeducation, correction of false beliefs, counseling to counteract barriers to hygienic practices, motivational enhancement, and behavioral skills training in hygiene practices
  Arms: Skin and Needle Hygiene Intervention
Other: No intervention - assessment-only condition — No intervention is assigned in this condition
  Arms: Assessment-Only Condition

SUMMARY:
The purpose of this study is to develop and test an intervention to reduce bacterial and viral infections among injection drug users.

DETAILED DESCRIPTION:
Injection drug use (IDU) is a major public health problem that is associated with a host of medical complications, including blood-borne viral disease (e.g., HIV, Hepatitis C) and bacterial infections (e.g., skin abscesses, endocarditis), that often result from high-risk drug injection practices. There are no current interventions designed to reduce bacterial infections among IDUs, despite high rates of infection.

The objective of this study is to develop and test the efficacy of a skin and needle hygiene intervention for IDUs to reduce practices associated with bacterial and viral infections. In the first phase of the study, focus group interviews were conducted to determine key areas of emphasis for an intervention with this population. An initial intervention was developed, pilot tested, and refined. The final 2-session intervention combines psychoeducation, skill-building, and motivational interviewing.

Following refinement of the intervention, a small randomized controlled trial (n = 60; 30 in each group) to examine the efficacy of the intervention compared to an assessment-only condition will be conducted. The goals of this two-year study are to: 1) reduce high-risk injection practices among active IDUs that lead to bacterial and viral infections, 2) improve skin and needle cleaning behavioral skills, and 3) increase skin cleaning prior to injection and reduce subcutaneous/intramuscular injection.

In addition to examining these goals over a six-month period, the acceptability and feasibility of the intervention will be examined.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* injection of heroin on at least three different days in the last week
* injection of heroin for at least three months
* visible track marks/puncture wounds from needles
* positive urine screen for heroin

Exclusion Criteria:

* currently exhibiting active psychotic symptoms
* cannot complete study assessments or the intervention
* cannot provide informed consent
* unable to provide names and contact information for at least two verifiable locator persons who will know where to find client
* plans to relocate from area or be jail over next six months
* have been in a Project Safe study in the last year
* report being pregnant or attempting to become pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Reduction in self-reported high-risk injection practices for bacterial infections (as measured through the Bacterial Infections Risk Scale for Injectors) | 1 month
Reduction in self-reported high-risk injection practices for bacterial infections (as measured through the Bacterial Infections Risk Scale for Injectors) | 6 months
Reduction in self-reported high-risk injection practices for HIV/HCV viral infections (as measured through the Risk Assessment Battery) | 1 month
Reduction in self-reported high-risk injection practices for HIV/HCV viral infections (as measured through the Risk Assessment Battery) | 6 months

SECONDARY OUTCOMES:
Improvement in skin and needle cleaning behavioral skills (as measured through Behavioral Skill Demonstration of Hand/Skin and Needle Cleaning) | 1 month
Increase in skin cleaning prior to injection and decrease in subcutaneous/intramuscular injection, as measured through Timeline Followback (TLFB) recall. | 1 month
Improvement in skin and needle cleaning behavioral skills (as measured through Behavioral Skill Demonstration of Hand/Skin and Needle Cleaning) | 6 months
Increase in skin cleaning prior to injection and decrease in subcutaneous/intramuscular injection, as measured through Timeline Followback (TLFB) recall. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Kristina T Phillips, Ph.D., Principal Investigator — University of Northern Colorado
Locations (1):
- Project Safe, University of Colorado, Denver, Colorado, United States